CLINICAL TRIAL: NCT01785420
Title: A Phase III Double Blind Randomized Placebo Controlled Study of Trastuzumab as Short Duration Preoperative Therapy in Patients With HER2-neu Positive Operable Breast Cancer
Brief Title: Pre Operative Trastuzumab in Operable Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dr Rajendra A. Badwe (Other Government)
Collaborators: Tata Memorial Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Dr Rajendra A. Badwe, Director and Professor , Surgical Oncology, Tata Memorial Hospital, Tata Memorial Hospital
Organization: Tata Memorial Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TMH Project-982
Record Dates: First submitted 2013-01-01; First posted 2013-02-07 (Estimated); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Carcinoma Breast Stage I; HER2 Positive Breast Cancer
Keywords: Pre-operative Trastuzumab Protocol
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug Trastuzumab (Experimental): A single dose of Trastuzumab (Herceptin, Hoffman La Roche) at 8 mg/Kg as a 90 minute infusion in 250 ml of normal saline, in the window period of 14 days (both days inclusive) prior to the planned date of surgery.
  Interventions: Drug: Trastuzumab
- Control (Placebo Comparator): A 90 minute intravenous infusion of saline as placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trastuzumab — A single dose of Trastuzumab (Herceptin, Hoffman La Roche) at 8 mg/Kg as a 90 minute infusion in 250 ml of normal saline, in the window period of 14 days (both days inclusive) prior to the planned date of surgery.
  Other Names: Herceptin
  Arms: Drug Trastuzumab
Drug: Placebo — A 90 minute intravenous infusion of saline as placebo
  Other Names: Normal saline
  Arms: Control

SUMMARY:
Background Information and Rationale:

Trastuzumab is a humanized monoclonal antibody that acts extracellularly on the erbB-2 receptor.Trastuzumab is a recombinant humanized IgG1 monoclonal antibody against the human epidermal growth factor receptor 2 (HER2/erbB-2),which has shown in both in vitro assays and in animals, to inhibit the proliferation of human tumour cells that overexpress erbB-2. Additionally, trastuzumab is a potent mediator of antibody-dependent cell-mediated cytotoxicity (ADCC). In vitro, trastuzumab-mediated ADCC has been shown to be preferentially exerted on erbB-2 overexpressing cancer cells compared with cancer cells that do not overexpress erbB-2. Trastuzumab has emerged as a widely accepted standard of care for erbB-2-positive disease. (Metastatic/ adjuvant/neoadjuvant.

Our current hypothesis suggests that the cells which are disseminated at the time of surgery will encounter an inhospitable environment which will be anti-HER in nature. Therefore combining the above mentioned streams of thought, we would like to assess the effect of a short pre-operative course of Trastuzumab on breast cancer relapse. The study is proposed in HER2 positive patients with operable breast cancer.

Objectives :

Primary:

The primary objective of the study is to see the effect of short duration of peri-operative Trastuzumab on disease-free survival in comparison in all patients

Secondary:

The safety of the pre-operative therapies including the early post operative morbidity

1. Overall survival (OS) in all patients and in pathologically node positive patients.
2. The level of circulating tumor cells (CTCs) in the peripheral blood assessed before starting pre-operative therapy and at the same time point in the control arm, level of CTCs 10 minutes prior to start of surgery, during surgery and 10 days after surgery on 40 consecutive consenting patients (20 in each arm). The levels of circulating chromatin will also be estimated at the same time points as CTC for these 40 patients.
3. Evaluation of the paraffin blocks for pTEN loss6-8 and p95ErbB2 truncated form of HER2 on 100 consecutive consenting patients (50 in each arm).9-11

Study Design :

This is phase 3, randomized Double blinded parallel group study of Trastuzumab in pre operative setting in operable breast cancer patients.

Approximately 1000 patients with Women with HER2neu positive, T1/T2/T3 and N0/N1. clinical T4 and/or N2 disease who are considered operable by the treating surgeon with histopathological diagnosis on core biopsies, will be included in the study. Patients with T4 or N2 (locally advanced and large operable for neo-adjuvant chemotherapy) will not be included. All node positive patients will receive single injection of Depot Inj. Progesterone 500 mg deep IM 4 -14 days prior to surgery

Patients will be stratified, before randomization for Tumor size, menopausal status, and affordability for Trastuzumab and centre of the study. These patients will then be randomized 1:1 to receive the following

Intervention arm: .A single dose of Trastuzumab (Herceptin, Hoffman La Roche) at 8 mg/Kg as a 90 minute intravenous infusion in 250 ml of normal saline, in the window period of 10-15 4 to 14 days (both days inclusive) prior to the planned date of surgery.

Control arm: A 90 minute intravenous infusion of saline as placebo

All patients will thereafter receive standard post-operative adjuvant therapy as per local institutional practice including hormonal therapy, chemotherapy and radiation therapy.

ELIGIBILITY:
Inclusion Criteria:a.

1. Female subjects aged 18 years or older.
2. Histologically and/or cytologically confirmed diagnosis of breast cancer. Clinical stages breast cancer: HER2 positive, T1 or T2 or T3, N0 or N1, resectable T4, or resectable N2, (all M0)
3. Documentation of erbB-2 gene amplification by FISH (as defined by a ratio >2.2) or chromogenic in situ hybridization (CISH, as defined by the manufacturer's kit instruction) or documentation of erbB-2-overexpression by IHC (defined as IHC3+, or IHC2+ with FISH or CISH confirmation) based on local laboratory.
4. LVEF within institutional range of normal as measured by MUGA or ECHO.
5. Screening laboratory values within the following parameters:

   1. Absolute neutrophil count (ANC) ≥1.5 x 109 /L (1500/mm3)
   2. Platelet count ≥100 x 109/L (100,000/mm3)
   3. Hemoglobin ≥9.0 g/dL (90 g/L)
   4. Serum creatinine ≤1.5 x upper limit of normal (ULN)
   5. Total bilirubin ≤1.5 x ULN (<3 ULN if Gilbert's disease) 6Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT)

      * 2.5 x ULN

Exclusion Criteria:

1. Bilateral breast cancer
2. Active uncontrolled cardiac disease, including cardiomyopathy, CHF (New York Heart Association [NYHA] functional classification of ≥3), unstable angina, and myocardial infarction (within 12 months of study entry).
3. Inadequately controlled hypertension (ie, systolic blood pressure [BP] > 180 mm Hg or diastolic BP > 100 mm Hg).
4. Family history of congenital long or short QT syndrome, Brugada syndrome or QT/QTc interval > 0.45 second or known history of QT/QTc prolongation or torsade de pointe (TdP).
5. Significant chronic gastrointestinal disorder with diarrhea as a major symptom (eg, Crohn's disease, malabsorption, or grade ≥2 diarrhea of any etiology at baseline).
6. Women who are pregnant, breast-feeding.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2013-05; Primary Completion 2025-04 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | up to 5 yrs
  Survival follow-up visits (or information Collected via telephone call) will be conducted approximately every 6 months (ie, 24 weeks) starting from the last day of primary (adjuvant) treatment.
  The subject will be called at clinic and will be carefully examined by a member of study team. A mammogram will be done every 18 months. If patient is symptomatic,additional investigations will be performed. Subject status as alive, alive with disease will be documented in the source file.

SECONDARY OUTCOMES:
Overall survival | Up to 5 yrs
  4.1.1. Overall survival (OS) in all patients and in pathologically node positive patients.
Circulating Tumour Cells in Peripheral Blood | 1. before starting pre-operative therapy and at the same time point in the control arm. 2. 10 minutes prior to start of surgery. 3. During surgery . 4. 10 days after surgery
4.1.3. Evaluation of the paraffin blocks for pTEN loss6-8 and p95ErbB2 truncated form of HER2 | upto 5 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Rajendra A Badwe, MS, Principal Investigator — Director and professor, Surgical Oncology
Locations (1):
- Tata Memorial Centre, Mumbai, India

REFERENCES:
- [Result] Burstein HJ, Sun Y, Dirix LY, Jiang Z, Paridaens R, Tan AR, Awada A, Ranade A, Jiao S, Schwartz G, Abbas R, Powell C, Turnbull K, Vermette J, Zacharchuk C, Badwe R. Neratinib, an irreversible ErbB receptor tyrosine kinase inhibitor, in patients with advanced ErbB2-positive breast cancer. J Clin Oncol. 2010 Mar 10;28(8):1301-7. doi: 10.1200/JCO.2009.25.8707. Epub 2010 Feb 8. PMID 20142587
- [Result] Badwe R, Hawaldar R, Parmar V, Nadkarni M, Shet T, Desai S, Gupta S, Jalali R, Vanmali V, Dikshit R, Mittra I. Single-injection depot progesterone before surgery and survival in women with operable breast cancer: a randomized controlled trial. J Clin Oncol. 2011 Jul 20;29(21):2845-51. doi: 10.1200/JCO.2010.33.0738. Epub 2011 Jun 13. PMID 21670457
- [Result] Ismail MS, Wynendaele W, Aerts JL, Paridaens R, Gaafar R, Shakankiry N, Khaled HM, Christiaens MR, Wildiers H, Omar S, Vandekerckhove P, Van Oosterom AT. Detection of micrometastatic disease and monitoring of perioperative tumor cell dissemination in primary operable breast cancer patients using real-time quantitative reverse transcription-PCR. Clin Cancer Res. 2004 Jan 1;10(1 Pt 1):196-201. doi: 10.1158/1078-0432.ccr-0515-2. PMID 14734470
- [Result] Nissen-Meyer R, Kjellgren K, Mansson B. Preliminary report from the Scandinavian adjuvant chemotherapy study group. Cancer Chemother Rep. 1971 Dec;55(5):561-6. No abstract available. PMID 4946080
- [Result] Nagata Y, Lan KH, Zhou X, Tan M, Esteva FJ, Sahin AA, Klos KS, Li P, Monia BP, Nguyen NT, Hortobagyi GN, Hung MC, Yu D. PTEN activation contributes to tumor inhibition by trastuzumab, and loss of PTEN predicts trastuzumab resistance in patients. Cancer Cell. 2004 Aug;6(2):117-27. doi: 10.1016/j.ccr.2004.06.022. PMID 15324695
- [Result] Depowski PL, Rosenthal SI, Ross JS. Loss of expression of the PTEN gene protein product is associated with poor outcome in breast cancer. Mod Pathol. 2001 Jul;14(7):672-6. doi: 10.1038/modpathol.3880371. PMID 11454999
- [Result] Fujita T, Doihara H, Kawasaki K, Takabatake D, Takahashi H, Washio K, Tsukuda K, Ogasawara Y, Shimizu N. PTEN activity could be a predictive marker of trastuzumab efficacy in the treatment of ErbB2-overexpressing breast cancer. Br J Cancer. 2006 Jan 30;94(2):247-52. doi: 10.1038/sj.bjc.6602926. PMID 16404430
- [Result] Saez R, Molina MA, Ramsey EE, Rojo F, Keenan EJ, Albanell J, Lluch A, Garcia-Conde J, Baselga J, Clinton GM. p95HER-2 predicts worse outcome in patients with HER-2-positive breast cancer. Clin Cancer Res. 2006 Jan 15;12(2):424-31. doi: 10.1158/1078-0432.CCR-05-1807. PMID 16428482
- [Result] Xia W, Liu LH, Ho P, Spector NL. Truncated ErbB2 receptor (p95ErbB2) is regulated by heregulin through heterodimer formation with ErbB3 yet remains sensitive to the dual EGFR/ErbB2 kinase inhibitor GW572016. Oncogene. 2004 Jan 22;23(3):646-53. doi: 10.1038/sj.onc.1207166. PMID 14737100
- [Result] Scaltriti M, Rojo F, Ocana A, Anido J, Guzman M, Cortes J, Di Cosimo S, Matias-Guiu X, Ramon y Cajal S, Arribas J, Baselga J. Expression of p95HER2, a truncated form of the HER2 receptor, and response to anti-HER2 therapies in breast cancer. J Natl Cancer Inst. 2007 Apr 18;99(8):628-38. doi: 10.1093/jnci/djk134. PMID 17440164
- [Result] Goldhirsch A, Glick JH, Gelber RD, Coates AS, Thurlimann B, Senn HJ; Panel members. Meeting highlights: international expert consensus on the primary therapy of early breast cancer 2005. Ann Oncol. 2005 Oct;16(10):1569-83. doi: 10.1093/annonc/mdi326. Epub 2005 Sep 7. PMID 16148022